CLINICAL TRIAL: NCT03836742
Title: Evaluation of Safety and Efficacy of a Regional Anticoagulation Protocol for Continuous Renal Replacement Therapies.
Brief Title: HEmoFiltration With Citric Acid Anticoagulation
Acronym: HEFCAA
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Romuald Lango, Prof. Romuald Lango, Medical University of Gdansk
Other Study IDs: NKBBN/539/2016-17
Record Dates: First submitted 2019-02-06; First posted 2019-02-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Acute Kidney Injury; Acute Kidney Failure; Renal Replacement Therapy; Hemofiltration
MeSH Terms: conditions — Acute Kidney Injury | interventions — Hemofiltration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HF RCA: Cardiovascular surgery patients treated with hemofiltration with regional citrate anticoagulation
  Interventions: Procedure: Hemofiltration with regional citrate anticoagulation

INTERVENTIONS:
Procedure: Hemofiltration with regional citrate anticoagulation — To reduce risk of metabolic alkalosis during hemofiltration treatment, ACD-A citrate solution was proposed instead of most commonly used trisodium citrate solution and relatively low target citrate concentration (2.8 mmol/L) was adopted. In case of pH increase above 7.5 or bicarbonate concentration above 40 mmol/L filtrate flow was decreased from initial 35 ml/kg/hour down to 25 ml/kg/hour which reduced bicarbonate delivery by 25%. If metabolic alkalosis persisted, the second step involved reduction of blood flow from initial 5 times down to 4 times filtrate flow, which reduced citrate flow by the same factor.

SUMMARY:
Prospective observational study of all consecutive cardio-vascular surgical patients treated with post-dilution hemofiltration with regional citrate anticoagulation as first-choice anticoagulation method. The filter life-span was assessed in the context of postoperative cardiac surgical antithrombotic prophylaxis. Reasons for termination of hemofiltration sessions were assessed. The second aim of this study was to assess the influence ACD-A based anticoagulation protocol on acid-base and ion homeostasis in cardiac surgical patients with acute renal failure.

DETAILED DESCRIPTION:
All consecutive cardio-vascular surgery patients treated with post-dilution hemofiltration with regional citrate anticoagulation (HF RCA) from August 2015 through November 2017 were included to prospective audit. Indication to hemofiltration treatment was based on clinical assessment of patients renal function and clinical status by attending physician and conformed conventional indications to renal replacement therapy (RRT) in intensive care unit (ICU). Severe chronic liver disease or acute liver injury with INR > 2 and refractory shock with lactate increasing above 8 mmol/L were considered as contraindication to RCA.

Initially set blood flow was 5 times higher than filtrate flow, which makes filtration fraction of 20%. To reduce the risk of metabolic alkalosis, ACD-A citrate solution was proposed instead of most commonly used trisodium citrate solution, and relatively low target citrate concentration (2.8 mmol/L) was adopted. In case of pH increase above 7.5 or bicarbonate concentration above 40 mmol/L filtrate flow was decreased from initial 35 ml/kg/hour down to 25 ml/kg/hour which should reduce bicarbonate synthesis by 25%. If metabolic alkalosis persisted, the second step involved reduction of blood flow from initial 5 times down to 4 times filtrate flow, which reduced citrate flow by the same factor.

In order to avoid hypomagnesemia resulting from magnesium binding to citrate, and its removal with ultrafiltrate not balanced with magnesium content in replacement fluid, the original protocol was modified by connecting magnesium sulfate solution 2g/50 ml 0.9% NaCl at the flow 1 mL/hour.

All sessions stopped due to patients death before 48 hours of HF treatment were excluded from the analysis. Similarly, all cases where hemofiltration session was stopped before 48 hours of treatment due to organizational reasons, recovery of renal function, change of therapy, and when patients were treated with heparin infusion due to surgical indications were excluded from further circuit survival analysis.

Blood gas parameters together with pH, bicarbonate concentration, Na, Cl, K, Ca, hemoglobin concentration, hematocrit, lactate, and anion gap were analyzed every 6 hours. Post filter ionized calcium concentration was not assessed. Serum phosphate, magnesium and total calcium was assessed every 24 hours during hemofiltration treatment with RCA.

ELIGIBILITY:
Inclusion Criteria:

* cardiac and vascular surgery patients treated with continuous hemofiltration with regional citrate anticoagulation

Exclusion Criteria:

* severe chronic liver disease, acute liver injury with INR > 2, and refractory shock with lactate increasing above 8 mmol/L

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive cardio-vascular surgery patients treated with post-dilution hemofiltration with regional citrate anticoagulation from August 2015 through November 2017
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Hemofiltration circuit survival time | up to 120 hours from the beginning of hemofiltration session
  in hours
Incidence of metabolic alkalosis | From the beginning of hemofiltration session until 6 hours after its end
  Arterial blood pH>7.5 or BE > 40 mmol/L
Incidence of hypernatremia and hyponatremia | From the beginning of hemofiltration session until 6 hours after its end
  Incidence of hypernatremia> 150 mmol/L and hyponatremia < 130 mmol/L in arterial blood sample

SECONDARY OUTCOMES:
Incidence of citrate accumulation | From the beginning of hemofiltration session until 24 hours after its end
  Incidence of total to ionized calcium ratio > 2,5 in arterial blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Romuald Lango, Gdansk, Polska, Poland

IPD SHARING:
Plan to Share IPD: No
No IPD are to be shared with other researcher

REFERENCES:
- [Background] Kirwan CJ, Hutchison R, Ghabina S, Schwarze S, Beane A, Ramsay S, Thompson E, Prowle JR. Implementation of a Simplified Regional Citrate Anticoagulation Protocol for Post-Dilution Continuous Hemofiltration Using a Bicarbonate Buffered, Calcium Containing Replacement Solution. Blood Purif. 2016;42(4):349-355. doi: 10.1159/000452755. Epub 2016 Nov 19. PMID 27866200